CLINICAL TRIAL: NCT01435486
Title: Caffeine Citrate for the Treatment of Apnea Associated With Bronchiolitis in Young Infants: A Randomized, Double Blind, Controlled Trial (RCT)
Brief Title: Caffeine Citrate for the Treatment of Apnea Associated With Bronchiolitis in Young Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: #11146/11
Record Dates: First submitted 2011-09-08; First posted 2011-09-16 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2014-05

CONDITIONS: Bronchiolitis; Apnea; Caffeine
Keywords: caffeine; apnea; bronchiolitis
MeSH Terms: conditions — Bronchiolitis; Apnea | interventions — caffeine citrate; Saline Solution; JPT1 protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- caffeine Citrate (Active Comparator)
  Interventions: Drug: Caffeine citrate
- Normal saline (Placebo Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Caffeine citrate — Single stat dose (25 mg per kilogram of body weight) of intravenous caffeine citrate (25mg caffeine citrate equal to 12.5mg caffeine base).
  Other Names: arm 1
  Arms: caffeine Citrate
Drug: Normal saline — Placebo with an equivalent volume of normal saline.
  Other Names: arm2
  Arms: Normal saline

SUMMARY:
Viral bronchiolitis is the most common lower respiratory tract infection of infancy. Apnea is a complication of bronchiolitis, reported in 16 - 21% of cases. Caffeine, a trimethylxanthine, acts as an antagonist to endogenous adenosine and a potent central nervous system stimulant. In apnea of prematurity, caffeine is believed to work by increasing central respiratory drive.

Infants ≤4 months of age, presenting to pediatric emergency center Al-Sadd, from September 2011 to May 2014, with a diagnosis of viral bronchiolitis associated with apnea.

A randomized, double-blind, controlled trial with a sample size of 45 patients per group

Data Collection methods, instruments used measurements:

Randomization:

In the emergency department, the patients will be assigned to either one of the two treatments using a computer-generated randomized numbers in a 1:1 ratio. Pharmacy will prepare sequential sealed vials containing the experimental drugs. Randomization code will be revealed only after all patients completed the study. The medical team in addition to the patients will be blinded to the medication delivered. There will be no detectable difference in the color, smell of the two study treatments.

Guardians or parents of eligible infants will be approached regarding the study, explaining the purpose and the treatment modalities. Patients will be included after obtaining a verbal and written consent.

Study Intervention:

Treatment 1: Single stat dose (25 mg per kilogram of body weight) of intravenous caffeine citrate (25mg caffeine citrate equal to 12.5mg caffeine base).

Treatment 2: Placebo with an equivalent volume of normal saline. Calculated study medications will be diluted with Dextrose 5% in Water to 20 ml and will be given intravenous over 30 minutes using syringe infusion pump.

After random assignment, eligible infants will receive one of the study treatments. Non-pharmacological therapies may be used as necessary to control apnea. Antibiotics and antipyretics may be used as per the discretion of the treating physician.

After stabilization of patients as usually done in Pediatric Emergency Center , patients will be admitted to pediatric intensive care unit (PICU) for further monitoring monitoring when indicated.

DETAILED DESCRIPTION:
Study area/setting:

Pediatric emergency center Al-Sadd, (PEC) is the main pediatric emergency centre in the state of Qatar with approximately 200,000 visits annually. It has a capacity of 42 observation beds providing most of the inpatient facilities except for intensive care monitoring. Patients admitted to the Pediatric Emergency Center are managed there until discharged home unless an Intensive Care Unit admission is required.

Study Subjects:

* Inclusion criteria: Infants ≤4 months of age, presenting to pediatric emergency center Al-Sadd, from September 2011 to May 2014, with a diagnosis of viral bronchiolitis associated with apnea.
* Exclusion criteria:

  * Hypersensitivity to caffeine.
  * Patients on caffeine treatment.
  * Cardiovascular congenital abnormalities.
  * Infants with a previous diagnosis of gastroesophageal reflux disease.
  * Hypoglycemia and/or electrolytes disorders.
  * Suspected sepsis.
  * Seizure disorders.
  * Inborn errors of metabolism.
  * Renal and/or hepatic impairment.
  * Major congenital anomalies of the upper and lower respiratory tract (severe tracheomalacia, trachea-esophageal fistula, diaphragmatic hernia, congenital lobar emphysema, congenital cystic adenomatoid malformation).

Study Design: A randomized, double-blind, controlled trial.

Sample Size:

In a retrospective chart review for all patients admitted to our institutions PICU/step-down unit with bronchiolitis associated with apnea in 2010, 87 patients were identified, 52 patients (60%) were apnea free after 12 hours from admission. To enable detection of a 50% improvement for the investigated group in resolution of apnea after 12 hours with 90% power and two sided alpha= 0.05, we estimated 42 patients per group is required. To compensate for dropouts, we planned to recruit 90 patients altogether.

Data Collection methods, instruments used measurements:

Randomization:

In the emergency department, the patients will be assigned to either one of the two treatments using a computer-generated randomized numbers in a 1:1 ratio. Pharmacy will prepare sequential sealed vials containing the experimental drugs. Randomization code will be revealed only after all patients completed the study. The medical team in addition to the patients will be blinded to the medication delivered. There will be no detectable difference in the color, smell of the two study treatments.

Guardians or parents of eligible infants will be approached regarding the study, explaining the purpose and the treatment modalities. Patients will be included after obtaining a verbal and written consent.

Study Intervention:

Treatment 1: Single stat dose (25 mg per kilogram of body weight) of intravenous caffeine citrate (25mg caffeine citrate equal to 12.5mg caffeine base).

Treatment 2: Placebo with an equivalent volume of normal saline.

Calculated study medications will be diluted with D5W to 20 ml and will be given intravenous over 30 minutes using syringe infusion pump.

After random assignment, eligible infants will receive one of the study treatments. Non-pharmacologic therapies such as supplemental oxygen, non invasive respiratory support, endotracheal intubation and mechanical ventilation may be used as necessary to control apnea. Antibiotics and antipyretics may be used as per the discretion of the treating physician.

After stabilization of patients as usually done in pediatric emergency center , patients will be admitted to Pediatric Intensive Care Unit for further monitoring when indicated.

ELIGIBILITY:
Inclusion Criteria:

* Infants ≤4 months of age, presenting to pediatric emergency center Al-Sadd, from September 2011 to May 2014, with a diagnosis of viral bronchiolitis associated with apnea.

Exclusion Criteria:

* Hypersensitivity to caffeine.
* Patients on caffeine treatment.
* Cardiovascular congenital abnormalities.
* Infants with a previous diagnosis of gastroesophageal reflux disease.
* Hypoglycemia and/or electrolytes disorders.
* Suspected sepsis.
* Seizure disorders.
* Inborn errors of metabolism.
* Renal and/or hepatic impairment.
* Major congenital anomalies of the upper and lower respiratory tract (severe tracheomalacia, trachea-esophageal fistula, diaphragmatic hernia, congenital lobar emphysema, congenital cystic adenomatoid malformation).

Ages: 1 Day to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2011-11; Primary Completion 2014-05 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
The primary efficacy outcome in this double-blinded study was the time until last apnea episode in both groups. | 2 year 8 mongths

SECONDARY OUTCOMES:
The proportion of patients with apnea resolution at 12 hours in both groups, | 2 year and 8 months
The frequency of apnea in the first 24, 48 and 72 hours after medication administration for both arms | 2 year and 8 months
The duration of apnea in the first 24, 48, and 72 hours after medication administration for both arms | 2 year and 8 months
Invasive and non-invasive respiratory support needed in both groups. | 2 year 8 months
The length of oxygen therapy needed in both groups. | 2 year 8 months
The time until feeding was tolerated in both groups. | 2 year 8 months
The length of PICU/step-down unit stay in both groups. | 2 year 8 months
The overall length of hospital stay in both groups. | 2 year 8 months
Spot heart rate in both groups was compared every 4 hours from enrollment for up to three days. | 2 year 8 months
  As a safety measure, spot heart rate was compared every 4 hours from enrollment for up to three days.

CONTACTS AND LOCATIONS:
Overall Officials: dr. Khalid Al-ansari, MD,FAAP, Principal Investigator — consultant pediatric emergency
Locations (1):
- Pediatric emergency center, Hamad Medical Corporation, Doha, Baladīyat ad Dawḩah, Qatar

REFERENCES:
- [Derived] Alansari K, Toaimah FH, Khalafalla H, El Tatawy LA, Davidson BL, Ahmed W. Caffeine for the Treatment of Apnea in Bronchiolitis: A Randomized Trial. J Pediatr. 2016 Oct;177:204-211.e3. doi: 10.1016/j.jpeds.2016.04.060. Epub 2016 May 14. PMID 27189681